CLINICAL TRIAL: NCT00412841
Title: AVN Prevention With Lipitor in Lupus Erythematosus APLLE Trial
Brief Title: Atorvastatin to Prevent Avascular Necrosis of Bone in Steroid Treated Exacerbated Systemic Lupus Erythematosus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-8795
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2018-11-23 (Actual); Status verified 2018-10

CONDITIONS: Avascular Necrosis
Keywords: Avascular Necrosis; Lipitor; SLE
MeSH Terms: conditions — Osteonecrosis | interventions — Atorvastatin; Magnetic Resonance Spectroscopy; Phlebotomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atorvastatin (Experimental): Atorvastatin 40mg
  Interventions: Drug: Atorvastatin; Procedure: MRI, Venipuncture
- Placebo (Placebo Comparator): Tablets identical to atorvastatin 40mg
  Interventions: Procedure: MRI, Venipuncture; Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 40mg vs placebo 40mg daily
  Other Names: Atorvasatatin 40mg vs Placebo
  Arms: Atorvastatin
Procedure: MRI, Venipuncture — MRIs done baseline, four and nine months
  Other Names: MRI at baseline, 4 months and 9 months
Drug: Placebo — Tablets identical to atorvastatin 40mg
  Arms: Placebo

SUMMARY:
This study uses the cholesterol lowering drug atorvastatin, also known as lipitor, to show reduction of avascular necrosis in steroid treated lupus patients. Avascular necrosis is a disease resulting from the loss of blood supply to the bones which can cause the bone to collapse. The collapse of bone may require a surgical replacement of the joint and can be disabling for life. Avascular necrosis is presently not preventable but research has shown that lipid lowering drugs such as lipitor can reduce or prevent avascular necrosis in animals. We therefore hypothesize that lipitor will reduce the incidence of avascular necrosis in lupus patients taking high dose steroids.

DETAILED DESCRIPTION:
If you have started on prednisone 30mg or greater and expect to be on it for greater than two weeks you may be a candidate for the study. Also, you would need to be enrolled in the study within three days of starting prednisone. If you are eligible you will receive lipitor 40mg per day or pills which look exactly like lipitor but do not contain any medication (called placebo). During the time of the study, you will not know if you are taking lipitor or the placebo. The period of time that you will receive lipitor or placebo is 9 months and you must be willing to return for 5 follow up visits during this time which include blood tests, physical exams and 3 MRI studies of the hips, knees and ankles.

ELIGIBILITY:
Inclusion Criteria:

* All individuals must fulfill 4 of the revised criteria of the American College of Rheumatology for SLE
* Patient started on corticosteroids at a dose of at least .5mg/kg for an interval greater than two weeks
* To be able to come for all follow-up visits for nine months
* No contraindications to undergoing MRI
* Age 18-75 years

Exclusion Criteria:

* Evidence of liver disease, not secondary to active lupus, or liver enzyme greater than 2x normal
* Elevated CPK at baseline
* Pregnancy or Lactating
* Allergy to a statin
* Current or recent use of a statin within 3 months

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2002-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard M Belmont, M.D., Principal Investigator — The New York University Hospital for Joint Diseases
Locations (1):
- The New York University Hospital For Joint Diseases, New York, New York, United States

REFERENCES:
- [Background] Belmont HM, Lydon E. Avascular necrosis prevention with lipitor in lupus erythematosus. Lupus. 2005;14(10):869-70. doi: 10.1191/0961203305lu2189xx. No abstract available. PMID 16302686

RESULTS

PARTICIPANT FLOW:
Groups:
- Atorvastatin: 40 mg
Period: Overall Study
Arm/Group | Atorvastatin | Placebo
Started | 22 | 21
Completed | 12 | 16
Not Completed | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin | Placebo | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 21 | 43
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 35 [18 to 58] | 35 [20 to 57] | 35 [18 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 22 | 21 | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With AVN After 9 Months
Time Frame: 9 months
Measure: Number; unit: participants
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 22 | 21
participants | 12 | 16

2. Secondary Outcome: Number of Participants With AVN After 4 Months
Time Frame: 4 months
Measure: Number; unit: participants
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 22 | 21
participants | 14 | 19

3. Secondary Outcome: To Determine if Atorvastatin is Effective in Lowering Serum Lipid Levels Chol, TG, HDL, & LDL in SLE Patients
Time Frame: 6 years
Population: Study Terminated. No data available for analysis. Secondary Outcome measure was not included in analysis.
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: To Determine if Atorvastatin Has an Anti-inflammatory Effect in Active SLE That Reduces Biological Markers of the Inflammatory Process (ESR, Hs-CRP) and Reduces Disease Activity Assessed by Serology (C3, C4, Anti-dsDNA) or Clinical Instrument (SLEDAI)
Time Frame: 6 years
Population: Study Terminated. No data available for analysis. Secondary Outcome measure was not included in analysis.
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Placebo: Placebo
Arm/Group | Atorvastatin | Placebo
Serious Adverse Events (participants affected / at risk) | 4/22 | 13/21
Other Adverse Events (participants affected / at risk) | 0/22 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin (N=22) | Placebo (N=21)
Fever of unknown origin (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fever, dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Elevated CPK (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Asystolic arrest (Cardiac disorders) | 0 (0) | 1 (1)
candida esophagitis (Infections and infestations) | 0 (0) | 1 (1)
elevated LFTS (Gastrointestinal disorders) | 0 (0) | 1 (1)
herpes zoster (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
pustular psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
UTI (Renal and urinary disorders) | 0 (0) | 1 (1)
vaginal candidiasis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
lung cancer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
tooth abscess (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No